CLINICAL TRIAL: NCT05623137
Title: Transcutaneous Electrical Nerve Stimulation (TENS) Over Acupoints (Acu-TENS) for Improving Sleep Quality, Cognitive Function, Motor Function and in Post-stroke Patients
Brief Title: Acu-TENS to Improve the Sleep Quality in People with Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022ShamayAcu-tens_Stroke
Record Dates: First submitted 2022-11-07; First posted 2022-11-21 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: AcuTENS; Sleep Quality; Stroke
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant
Masking Description: Due to the nature of the treatments, only the participants will be blinded to the objectives of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acu-TENS+SHP (Experimental): The 120z Dual-Channel TENS Unit (ECS300A; Neurotrac, Verity Medical LTD, Ireland) will be used to stimulate the selected acupoints. The electrode will be placed over the acupoints and connected to the TENS stimulator. The stimulation frequency will be set at 100 Hz with a pulse width of 0.2 ms. Participants will also receive a set of instructions relating to SHP. SHP is a set of instructions designed to help with sleep and promote healthy sleeping habits. Participants will be instructed to read the guide after the baseline assessment (T0).
  Interventions: Device: Acu-TENS; Other: SHP
- Sham Acu-TENS+SHP (Sham Comparator): Participants will receive similar treatment as Acu-TENS groups via identical-looking TENS devices with the electrical circuit disconnected.Participants will also receive a set of instructions relating to SHP. SHP is a set of instructions designed to help with sleep and promote healthy sleeping habits. Participants will be instructed to read the guide after the baseline assessment (T0).
  Interventions: Device: Sham Acu-TENS; Other: SHP

INTERVENTIONS:
Device: Acu-TENS — A dual-channel TENS stimulator will be used (ECS300A; Neurotrac, Verity Medical LTD, Ireland). Electrodes will be placed over selected acupoints (i.e., bilateral Sanyinjiao (SP6), Neiguan (PC6), Shenmen (HT7), Hegu (LI4), Zusanli (ST36) and Quchi (LI11)) and connected to the TENS stimulator. These acupoints are selected according to the traditional Chinese medicine and results of previous studies. The stimulation will be lasted 30-min for each session. The frequency of the stimulation parameter's waveform will be set to 100 Hz and the square pulses will be set to 0.2-ms. The intensity of the stimulation will be below motor threshold and lower than the intolerable level, and hence, participants will feel a pleasant and mild aching sensation.
  Arms: Acu-TENS+SHP
Device: Sham Acu-TENS — A dual-channel TENS stimulator will be used (ITO Physiotherapy & Rehabilitation, Co, Ltd, Tokyo, Japan). Electrodes will be placed over selected acupoints (i.e., bilateral Sanyinjiao (SP6), Neiguan (PC6), Shenmen (HT7), Hegu (LI4), Zusanli (ST36) and Quchi (LI11)) and connected to the TENS stimulator. These acupoints are selected according to the traditional Chinese medicine and results of previous studies. The stimulation will be lasted 30-min for each session. The frequency of the stimulation parameter's waveform will be set to 100 Hz and the square pulses will be set to 0.2-ms. The intensity of the stimulation will be below motor threshold and lower than the intolerable level, and hence, participants will feel a pleasant and mild aching sensation.
  Arms: Sham Acu-TENS+SHP
Other: SHP — SHP is a set of instructions designed to help with sleep and promote healthy sleeping habits. The sleep guide contains information on how much sleep is needed by every individual daily, factors that could affect sleep, and risk factors for sleep disorders. It also contains information on the types of sleep disorders, delayed sleep syndrome, insomnia-producing behavior that could affect sleep quality, and suggestions for inducing sleep. The participants will be instructed to read the guide after the baseline assessment (T0). Those instructions will be reinforced by the research practitioner after each treatment session, in order to maintain the healthy sleeping habits.

SUMMARY:
Post-stroke sleep disorder and motor/cognitive dysfunction are common complications that affect the quality of life of older patients. The proposed study investigates the effects of an acupuncture-like method applied to six bilateral acupoints on sleep quality, motor function and cognition in older adults with chronic stroke. The study will be a single-blind (i.e., only patients will be blinded about the research purpose) randomized controlled trial (i.e., patients receiving the treatment is chosen at random) with a pre-mid-post follow-up design and involve two parallel groups of post-stroke survivors (aged > 55 years) diagnosed with insomnia. Participants will be randomly allocated in a 1:1 radio to two independent groups, i.e., a treatment group or placebo group, namely a transcutaneous electrical nerve stimulation placed on acupoints (Acu-TENS) or a placebo group. The Acu-TENS group will receive a 6-week treatment that includes a 30-minute Acu-TENS + sleep hygiene program (SHP) twice a week. The placebo group will receive sham Acu-TENS (i.e., devices with the electrical circuit disconnected) + SHP with the same frequency as the Acu-TENS group. The selected acupoints will be bilateral Hegu (LI4), Quchi (LI11), Neiguan (PC6), Shenmen (HT7) on the arm and Sanyinjiao (SP6) and Zusanli (ST36) on the lower limb. The study's primary outcomes will be sleep quality measured by the device of ActiGraph and the self-report survey. The secondary outcomes will be motor function, measured by physical performance tests, cognition, measured by computer battery, and quality of life, measured by the self-report survey. All outcomes will be measured at the baseline assessment (before the treatment), mid-term assessment (after the three weeks treatment), post-treatment assessment (after the six-week treatment), and follow-up assessment (two weeks after the treatment ended). It is hypothesized that the Acu-TENS + SHP treatment will better alleviate insomnia, improve cognition and motor function in participants than the sham Acu-TENS + SHP treatment.

DETAILED DESCRIPTION:
The proposed study investigates the effects of non-invasive acupuncture techniques (i.e. transcutaneous electrical nerve stimulation at acupoints; Acu-TENS) applied to six selected bilateral acupoints on sleep quality, motor function and cognition in older adult participants with chronic stroke. This proposed project aims to investigate the effectiveness of Acu-TENS + sleep hygiene program (SHP), compare with placebo-stimulation +SHP on sleep quality, motor function and cognition, and quality of life of older adults with chronic stroke.

Impact:

1. Practical significance: The proposed clinical-based randomized controlled trial will rigorously investigate the effects of Acu-TENS applied to selected acupoints on sleep quality, motor function, cognition, and quality of life in older adults with chronic stroke. The results of this study will shed light on the effectiveness of this non-invasive acupuncture treatment for treating insomnia and improving motor and cognition function in older adults with chronic stroke. This will help healthcare professionals treat this highly prevalent disorder for which effective treatments are currently lacking.
2. Scientific significance: The proposed study will be the first to investigate the effects of Acu-TENS on elderly patients with post-stroke insomnia. The objective measures used in the rigorously designed study will generate high-quality data and produce rigorous results.

ELIGIBILITY:
Inclusion Criteria:

* aged between 55 and 85 yrs;
* diagnosed with stroke by magnetic resonance imaging or computed tomographic scan longer than one year;
* able to walk 6-m independently;
* scored ≥18 but less or equal than 27 in mini-mental state examination (MMSE);
* self-reported poor sleep quality (PSQI, scores ≥ 6) in the past four weeks.

Exclusion Criteria:

* have a cardiac pacemaker;
* have a severe disease that precludes the receipt of Acu-TENS;
* are taking medication that may affect measured outcomes;
* have skin lesions, infection, or inflammation near selected acupoints;
* are participating in other drug/treatment programs.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index (PSQI) | T0, baseline
  The subjective sleep quality will be assessed by the Pittsburgh sleep quality index. It has been used in both research and clinical settings to evaluate sleep quality and screen for sleep disturbances. The scores ranges from 0 to 21. A higher score means a lower sleep quality, with a score ≥ 6 as the cut-off value for poor sleep quality. The Chinese version will be used in the proposed study.
Pittsburgh sleep quality index (PSQI) | T1, mid (2th week)
  The subjective sleep quality will be assessed by the Pittsburgh sleep quality index. It has been used in both research and clinical settings to evaluate sleep quality and screen for sleep disturbances. The scores ranges from 0 to 21. A higher score means a lower sleep quality, with a score ≥ 6 as the cut-off value for poor sleep quality. The Chinese version will be used in the proposed study.
Pittsburgh sleep quality index (PSQI) | T2, post (4th week)
  The subjective sleep quality will be assessed by the Pittsburgh sleep quality index. It has been used in both research and clinical settings to evaluate sleep quality and screen for sleep disturbances. The scores ranges from 0 to 21. A higher score means a lower sleep quality, with a score ≥ 6 as the cut-off value for poor sleep quality. The Chinese version will be used in the proposed study.
Pittsburgh sleep quality index (PSQI) | T3, follow-up(6th week)
  The subjective sleep quality will be assessed by the Pittsburgh sleep quality index. It has been used in both research and clinical settings to evaluate sleep quality and screen for sleep disturbances. The scores ranges from 0 to 21. A higher score means a lower sleep quality, with a score ≥ 6 as the cut-off value for poor sleep quality. The Chinese version will be used in the proposed study.
Total sleep time | T0, baseline
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants' total sleep time (total time asleep from sleep onset to waking). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T2, T3). The validity of this assessment was confirmed in previous research.
Total sleep time | T2, post (4th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants' total sleep time (total time asleep from sleep onset to waking). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T2, T3). The validity of this assessment was confirmed in previous research.
Total sleep time | T3, follow-up(6th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants' total sleep time (total time asleep from sleep onset to waking). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T2, T3). The validity of this assessment was confirmed in previous research.
Sleep efficiency | T0, baseline
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants' sleep efficiency (percentage of total time in bed trying to sleep). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T2, T3). The validity of this assessment was confirmed in previous research.
Sleep efficiency | T2, post (4th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants' sleep efficiency (percentage of total time in bed trying to sleep). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T2, T3). The validity of this assessment was confirmed in previous research.
Sleep efficiency | T3, follow-up(6th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants' sleep efficiency (percentage of total time in bed trying to sleep). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T2, T3). The validity of this assessment was confirmed in previous research.
Sleep onset latency | T0, baseline
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants'sleep onset latency (time to fall asleep). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T2, T3). The validity of this assessment was confirmed in previous research.
Sleep onset latency | T2, post (4th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants'sleep onset latency (time to fall asleep). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T2, T3). The validity of this assessment was confirmed in previous research.
Sleep onset latency | T3, follow-up(6th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants'sleep onset latency (time to fall asleep). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T2, T3). The validity of this assessment was confirmed in previous research.
Time awake after sleep onset | T0, baseline
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants'time awake after sleep onset (total time awake from sleep onset to waking). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T2, T3). The validity of this assessment was confirmed in previous research.
Time awake after sleep onset | T2, post (4th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants'time awake after sleep onset (total time awake from sleep onset to waking). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T2, T3). The validity of this assessment was confirmed in previous research.
Time awake after sleep onset | T3, follow-up(6th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants'time awake after sleep onset (total time awake from sleep onset to waking). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T2, T3). The validity of this assessment was confirmed in previous research.
Insomnia severity index (ISI) | T0, baseline
  The subjective perception of the severity of insomnia will be assessed by Insomnia severity index. It comprises seven items measuring the severity of sleep-onset and sleep maintenance difficulties (both nocturnal and early-morning awakenings), satisfaction with the current sleep pattern, the adverse effects of insomnia on daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a scale from 0 to 4, and the total score ranges from 0 to 28. A higher score represents more severe insomnia. The Chinese version will be used in the proposed study.
Insomnia severity index (ISI) | T1, mid (2th week)
  The subjective perception of the severity of insomnia will be assessed by Insomnia severity index. It comprises seven items measuring the severity of sleep-onset and sleep maintenance difficulties (both nocturnal and early-morning awakenings), satisfaction with the current sleep pattern, the adverse effects of insomnia on daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a scale from 0 to 4, and the total score ranges from 0 to 28. A higher score represents more severe insomnia. The Chinese version will be used in the proposed study.
Insomnia severity index (ISI) | T2, post (4th week)
  The subjective perception of the severity of insomnia will be assessed by Insomnia severity index. It comprises seven items measuring the severity of sleep-onset and sleep maintenance difficulties (both nocturnal and early-morning awakenings), satisfaction with the current sleep pattern, the adverse effects of insomnia on daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a scale from 0 to 4, and the total score ranges from 0 to 28. A higher score represents more severe insomnia. The Chinese version will be used in the proposed study.
Insomnia severity index (ISI) | T3, follow-up(6th week)
  The subjective perception of the severity of insomnia will be assessed by Insomnia severity index. It comprises seven items measuring the severity of sleep-onset and sleep maintenance difficulties (both nocturnal and early-morning awakenings), satisfaction with the current sleep pattern, the adverse effects of insomnia on daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a scale from 0 to 4, and the total score ranges from 0 to 28. A higher score represents more severe insomnia. The Chinese version will be used in the proposed study.

SECONDARY OUTCOMES:
Stroop Color and Word Test | T0, baseline
  The ability to inhibit cognitive interference will be measured by the Stroop Color and Word Test. The Stroop Test consists of 3 subtasks. The first subtask shows color dots (green, blue, yellow, red) in random order. The second subtask shows the words (green, blue, red, yellow) in random order. The third task showed color words (green, blue, red, yellow) printed in a different ink color (i.e., the word blue printed in yellow ink). Participants are required to name the color of the ink as quickly as possible within 45 s in each task. The completion time and number of error is recorded in each task. The interference ratio of will be calculated as the completion time of the third task/the completion time of the first task. A higher interference score indicated poorer interference control.
Stroop Color and Word Test | T1, mid (2th week)
  The ability to inhibit cognitive interference will be measured by the Stroop Color and Word Test. The Stroop Test consists of 3 subtasks. The first subtask shows color dots (green, blue, yellow, red) in random order. The second subtask shows the words (green, blue, red, yellow) in random order. The third task showed color words (green, blue, red, yellow) printed in a different ink color (i.e., the word blue printed in yellow ink). Participants are required to name the color of the ink as quickly as possible within 45 s in each task. The completion time and number of error is recorded in each task. The interference ratio of will be calculated as the completion time of the third task/the completion time of the first task. A higher interference score indicated poorer interference control.
Stroop Color and Word Test | T2, post (4th week)
  The ability to inhibit cognitive interference will be measured by the Stroop Color and Word Test. The Stroop Test consists of 3 subtasks. The first subtask shows color dots (green, blue, yellow, red) in random order. The second subtask shows the words (green, blue, red, yellow) in random order. The third task showed color words (green, blue, red, yellow) printed in a different ink color (i.e., the word blue printed in yellow ink). Participants are required to name the color of the ink as quickly as possible within 45 s in each task. The completion time and number of error is recorded in each task. The interference ratio of will be calculated as the completion time of the third task/the completion time of the first task. A higher interference score indicated poorer interference control.
Stroop Color and Word Test | T3, follow-up(6th week)
  The ability to inhibit cognitive interference will be measured by the Stroop Color and Word Test. The Stroop Test consists of 3 subtasks. The first subtask shows color dots (green, blue, yellow, red) in random order. The second subtask shows the words (green, blue, red, yellow) in random order. The third task showed color words (green, blue, red, yellow) printed in a different ink color (i.e., the word blue printed in yellow ink). Participants are required to name the color of the ink as quickly as possible within 45 s in each task. The completion time and number of error is recorded in each task. The interference ratio of will be calculated as the completion time of the third task/the completion time of the first task. A higher interference score indicated poorer interference control.
Trail making test | T0, baseline
  The attention and cognitive flexibility will be assessed by trial making test. The test is divided into two parts: A and B. In part A, the circle is numbered (i.e., 1 to 25). The participants should draw lines in numeric order of the listed circle. In part B, the circles include both numbers (i.e., 1 to 13) and words (i.e., A to L); the participants should draw the lines in a specific sequence between number and word (i.e., 1 to A to 2 to B etc.). The test will be timed with a shorter time indicated the better performance. The test-retest reliability is good in stroke patients (ICC; 0.94 and 0.86 for Part A and Part B, respectively)
Trail making test | T1, mid (2th week)
  The attention and cognitive flexibility will be assessed by trial making test. The test is divided into two parts: A and B. In part A, the circle is numbered (i.e., 1 to 25). The participants should draw lines in numeric order of the listed circle. In part B, the circles include both numbers (i.e., 1 to 13) and words (i.e., A to L); the participants should draw the lines in a specific sequence between number and word (i.e., 1 to A to 2 to B etc.). The test will be timed with a shorter time indicated the better performance. The test-retest reliability is good in stroke patients (ICC; 0.94 and 0.86 for Part A and Part B, respectively)
Trail making test | T2, post (4th week)
  The attention and cognitive flexibility will be assessed by trial making test. The test is divided into two parts: A and B. In part A, the circle is numbered (i.e., 1 to 25). The participants should draw lines in numeric order of the listed circle. In part B, the circles include both numbers (i.e., 1 to 13) and words (i.e., A to L); the participants should draw the lines in a specific sequence between number and word (i.e., 1 to A to 2 to B etc.). The test will be timed with a shorter time indicated the better performance. The test-retest reliability is good in stroke patients (ICC; 0.94 and 0.86 for Part A and Part B, respectively)
Trail making test | T3, follow-up (6th week)
  The attention and cognitive flexibility will be assessed by trial making test. The test is divided into two parts: A and B. In part A, the circle is numbered (i.e., 1 to 25). The participants should draw lines in numeric order of the listed circle. In part B, the circles include both numbers (i.e., 1 to 13) and words (i.e., A to L); the participants should draw the lines in a specific sequence between number and word (i.e., 1 to A to 2 to B etc.). The test will be timed with a shorter time indicated the better performance. The test-retest reliability is good in stroke patients (ICC; 0.94 and 0.86 for Part A and Part B, respectively)
10-m walk test | T0, baseline
  The functional mobility will be assessed by the 10-m walk test. Participants will be instructed to walk without assistance for a 10-m distance in a solid flooring with a clear pathway. A mark at 2-m and 8-m will be placed. A stopwatch will be timed central 6-m to assess participants' acceleration and deceleration. It has shown good test-retested reliability in stroke patients.
10-m walk test | T1, mid (2th week)
  The functional mobility will be assessed by the 10-m walk test. Participants will be instructed to walk without assistance for a 10-m distance in a solid flooring with a clear pathway. A mark at 2-m and 8-m will be placed. A stopwatch will be timed central 6-m to assess participants' acceleration and deceleration. It has shown good test-retested reliability in stroke patients.
10-m walk test | T2, post (4th week)
  The functional mobility will be assessed by the 10-m walk test. Participants will be instructed to walk without assistance for a 10-m distance in a solid flooring with a clear pathway. A mark at 2-m and 8-m will be placed. A stopwatch will be timed central 6-m to assess participants' acceleration and deceleration. It has shown good test-retested reliability in stroke patients.
10-m walk test | T3, follow-up (6th week)
  The functional mobility will be assessed by the 10-m walk test. Participants will be instructed to walk without assistance for a 10-m distance in a solid flooring with a clear pathway. A mark at 2-m and 8-m will be placed. A stopwatch will be timed central 6-m to assess participants' acceleration and deceleration. It has shown good test-retested reliability in stroke patients.
Time up and go test | T0, baseline
  The walking mobility will be assessed by the Time up and go test. During the test, participants will be instructed to stand up from the chair, walk forward for 3-meter, turn around 180 degrees, walk back, and sit on the chair. The time taken to complete this task will be measured via stopwatch. The test has shown good test-retested reliability in stroke patients.
Time up and go test | T1, mid (2th week)
  The walking mobility will be assessed by the Time up and go test. During the test, participants will be instructed to stand up from the chair, walk forward for 3-meter, turn around 180 degrees, walk back, and sit on the chair. The time taken to complete this task will be measured via stopwatch. The test has shown good test-retested reliability in stroke patients.
Time up and go test | T2, post (4th week)
  The walking mobility will be assessed by the Time up and go test. During the test, participants will be instructed to stand up from the chair, walk forward for 3-meter, turn around 180 degrees, walk back, and sit on the chair. The time taken to complete this task will be measured via stopwatch. The test has shown good test-retested reliability in stroke patients.
Time up and go test | T3, follow-up (6th week)
  The walking mobility will be assessed by the Time up and go test. During the test, participants will be instructed to stand up from the chair, walk forward for 3-meter, turn around 180 degrees, walk back, and sit on the chair. The time taken to complete this task will be measured via stopwatch. The test has shown good test-retested reliability in stroke patients.
Lower limb muscle strength | T0, baseline
  The lower limb muscle strength of affected and unaffected ankle dorsiflexors and plantar flexors will be assessed by the hand-held dynamometer (Lafayette Hand-held Dynamometer Model 1165A, Lafayette Instrument Evaluation, Lafayette, Indiana, USA). The subjects will be asked to perform in the supine position. The hand-held dynamometer was positioned anteriorly or posteriorly over the heads of the first to fifth metatarsal bones to measure the strength of the ankle dorsiflexors and plantar flexors, respectively. Subjects were placed in the supine position and asked to perform the MIVC for 3 s. Each muscle group was tested twice by the same rater, with at least 30 s of rest between the two trials to reduce the effects of fatigue. The averages of the MIVC in kilograms were used in statistical analysis. The dynamometer used in the trials was shown to have excellent inter-rater reliability and test-retest reliability in community-dwelling older adults.
Lower limb muscle strength | T1, mid (2th week)
  The lower limb muscle strength of affected and unaffected ankle dorsiflexors and plantar flexors will be assessed by the hand-held dynamometer (Lafayette Hand-held Dynamometer Model 1165A, Lafayette Instrument Evaluation, Lafayette, Indiana, USA). The subjects will be asked to perform in the supine position. The hand-held dynamometer was positioned anteriorly or posteriorly over the heads of the first to fifth metatarsal bones to measure the strength of the ankle dorsiflexors and plantar flexors, respectively. Subjects were placed in the supine position and asked to perform the MIVC for 3 s. Each muscle group was tested twice by the same rater, with at least 30 s of rest between the two trials to reduce the effects of fatigue. The averages of the MIVC in kilograms were used in statistical analysis. The dynamometer used in the trials was shown to have excellent inter-rater reliability and test-retest reliability in community-dwelling older adults.
Lower limb muscle strength | T2, post (4th week)
  The lower limb muscle strength of affected and unaffected ankle dorsiflexors and plantar flexors will be assessed by the hand-held dynamometer (Lafayette Hand-held Dynamometer Model 1165A, Lafayette Instrument Evaluation, Lafayette, Indiana, USA). The subjects will be asked to perform in the supine position. The hand-held dynamometer was positioned anteriorly or posteriorly over the heads of the first to fifth metatarsal bones to measure the strength of the ankle dorsiflexors and plantar flexors, respectively. Subjects were placed in the supine position and asked to perform the MIVC for 3 s. Each muscle group was tested twice by the same rater, with at least 30 s of rest between the two trials to reduce the effects of fatigue. The averages of the MIVC in kilograms were used in statistical analysis. The dynamometer used in the trials was shown to have excellent inter-rater reliability and test-retest reliability in community-dwelling older adults.
Lower limb muscle strength | T3, follow-up (6th week)
  The lower limb muscle strength of affected and unaffected ankle dorsiflexors and plantar flexors will be assessed by the hand-held dynamometer (Lafayette Hand-held Dynamometer Model 1165A, Lafayette Instrument Evaluation, Lafayette, Indiana, USA). The subjects will be asked to perform in the supine position. The hand-held dynamometer was positioned anteriorly or posteriorly over the heads of the first to fifth metatarsal bones to measure the strength of the ankle dorsiflexors and plantar flexors, respectively. Subjects were placed in the supine position and asked to perform the MIVC for 3 s. Each muscle group was tested twice by the same rater, with at least 30 s of rest between the two trials to reduce the effects of fatigue. The averages of the MIVC in kilograms were used in statistical analysis. The dynamometer used in the trials was shown to have excellent inter-rater reliability and test-retest reliability in community-dwelling older adults.
The Fatigue Assessment Scale | T0, baseline
  The general fatigue will be assessed by The Fatigue Assessment Scale. It is a 10-item survey, of which 5 items assess physical fatigue and the remaining 5 items assess mental fatigue. The total score ranges from 10 to 50, and a total score ≥ 22 indicates fatigue. The translated Chinese version will be used in the proposed study.
The Fatigue Assessment Scale | T1, mid (2th week)
  The general fatigue will be assessed by The Fatigue Assessment Scale. It is a 10-item survey, of which 5 items assess physical fatigue and the remaining 5 items assess mental fatigue. The total score ranges from 10 to 50, and a total score ≥ 22 indicates fatigue. The translated Chinese version will be used in the proposed study.
The Fatigue Assessment Scale | T2, post (4th week)
  The general fatigue will be assessed by The Fatigue Assessment Scale. It is a 10-item survey, of which 5 items assess physical fatigue and the remaining 5 items assess mental fatigue. The total score ranges from 10 to 50, and a total score ≥ 22 indicates fatigue. The translated Chinese version will be used in the proposed study.
The Fatigue Assessment Scale | T3, follow-up (6th week)
  The general fatigue will be assessed by The Fatigue Assessment Scale. It is a 10-item survey, of which 5 items assess physical fatigue and the remaining 5 items assess mental fatigue. The total score ranges from 10 to 50, and a total score ≥ 22 indicates fatigue. The translated Chinese version will be used in the proposed study.
Depression Anxiety Stress Scale | T0, baseline
  Participants' mood will be measured by the Depression Anxiety Stress Scale, a 21-item survey that assesses depression, anxiety, and stress. Each index (i.e., depression, anxiety, and stress) comprises seven items. The scores ranges from 0 to 42. Higher score indicates more sever symptom. The reliability of this scale was confirmed in previous research.
Depression Anxiety Stress Scale | T1, mid (2th week)
  Participants' mood will be measured by the Depression Anxiety Stress Scale, a 21-item survey that assesses depression, anxiety, and stress. Each index (i.e., depression, anxiety, and stress) comprises seven items. The scores ranges from 0 to 42. Higher score indicates more sever symptom. The reliability of this scale was confirmed in previous research.
Depression Anxiety Stress Scale | T2, post (4th week)
  Participants' mood will be measured by the Depression Anxiety Stress Scale, a 21-item survey that assesses depression, anxiety, and stress. Each index (i.e., depression, anxiety, and stress) comprises seven items. The scores ranges from 0 to 42. Higher score indicates more sever symptom. The reliability of this scale was confirmed in previous research.
Depression Anxiety Stress Scale | T3, follow-up (6th week)
  Participants' mood will be measured by the Depression Anxiety Stress Scale, a 21-item survey that assesses depression, anxiety, and stress. Each index (i.e., depression, anxiety, and stress) comprises seven items. The scores ranges from 0 to 42. Higher score indicates more sever symptom. The reliability of this scale was confirmed in previous research.
Natural Oscillation Frequency | T0, baseline
  The Natural Oscillation Frequency will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Natural Oscillation Frequency | T1, mid (2th week)
  The Natural Oscillation Frequency will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Natural Oscillation Frequency | T2, post (4th week)
  The Natural Oscillation Frequency will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Natural Oscillation Frequency | T3, follow-up (6th week)
  The Natural Oscillation Frequency will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Health-related Quality of Life | T0, baseline
  The Health-related Quality of Life will be assessed by the 12-item Short-Form Survey (SF-12). This instrument contains eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The total score ranges from 0 to 100, with a higher score indicating better QoL.
Health-related Quality of Life | T1, mid (2th week)
  The Health-related Quality of Life will be assessed by the 12-item Short-Form Survey (SF-12). This instrument contains eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The total score ranges from 0 to 100, with a higher score indicating better QoL.
Health-related Quality of Life | T2, post (4th week)
  The Health-related Quality of Life will be assessed by the 12-item Short-Form Survey (SF-12). This instrument contains eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The total score ranges from 0 to 100, with a higher score indicating better QoL.
Health-related Quality of Life | T3, follow-up (6th week)
  The Health-related Quality of Life will be assessed by the 12-item Short-Form Survey (SF-12). This instrument contains eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The total score ranges from 0 to 100, with a higher score indicating better QoL.
Dynamic Stiffness | T0, baseline
  The Dynamic Stiffness will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Dynamic Stiffness | T1, mid (2th week)
  The Dynamic Stiffness will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Dynamic Stiffness | T2, post (4th week)
  The Dynamic Stiffness will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Dynamic Stiffness | T3, follow-up (6th week)
  The Dynamic Stiffness will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Logarithmic Decrement of natural oscillation | T0, baseline
  The Logarithmic Decrement of natural oscillation will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Logarithmic Decrement of natural oscillation | T1, mid (2th week)
  The Logarithmic Decrement of natural oscillation will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Logarithmic Decrement of natural oscillation | T2, post (4th week)
  The Logarithmic Decrement of natural oscillation will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Logarithmic Decrement of natural oscillation | T3, follow-up (6th week)
  The Logarithmic Decrement of natural oscillation will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Mechanical Stress Relaxation Time | T0, baseline
  The Mechanical Stress Relaxation Time will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Mechanical Stress Relaxation Time | T1, mid (2th week)
  The Mechanical Stress Relaxation Time will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Mechanical Stress Relaxation Time | T2, post (4th week)
  The Mechanical Stress Relaxation Time will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
Mechanical Stress Relaxation Time | T3, follow-up (6th week)
  The Mechanical Stress Relaxation Time will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
The Ratio of deformation and Relaxation time | T0, baseline
  The Ratio of deformation and Relaxation time will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
The Ratio of deformation and Relaxation time | T1, mid (2th week)
  The Ratio of deformation and Relaxation time will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
The Ratio of deformation and Relaxation time | T2, post (4th week)
  The Ratio of deformation and Relaxation time will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.
The Ratio of deformation and Relaxation time | T3, follow-up (6th week)
  The Ratio of deformation and Relaxation time will be used to assess the muscle stiffness. The muscle stiffness of the affected and unaffected lower limb will be assessed by a hand-held digit palpation device, MyotoPRO (Myoton AS, Tallinn, Estonia). The subject will be asked to perform in the sitting position with hip flexion 90°, knee flexion 90°. The standard probe was placed perpendicularly to the skin's surface of the affected and unaffected tibial anterior and medial gastrocnemius directly. An initial force was exerted; then, an additional mechanical force was applied to the subcutaneous tissue for 15 milliseconds, which induced muscle deformation. The resultant damped natural oscillations caused by the viscoelastic properties of the soft tissue were recorded using a built-in accelerometer at a sampling rate of 3200 Hz.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - The Hong Kong Polytechnic University, Hong Kong
  - The Hongkong Polytechnic University, Hong Kong